CLINICAL TRIAL: NCT00089856
Title: A Phase III Randomized, Open-Label Study of CG1940 and CG8711 Versus Docetaxel and Prednisone in Patients With Metastatic Hormone-Refractory Prostate Cancer Who Are Chemotherapy-Naïve
Brief Title: GVAX® Vaccine for Prostate Cancer vs Docetaxel & Prednisone in Patients With Metastatic Hormone-Refractory Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on futility analysis showing <30% chance of meeting primary endpoint.
Sponsor: Cell Genesys (Industry)
Responsible Party: Cell Genesys, Inc, Cell Genesys, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-0029; (VITAL-1)
Record Dates: First submitted 2004-08-16; First posted 2004-08-18 (Estimated); Last update posted 2008-11-05 (Estimated); Status verified 2008-11

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Metastatic; Hormone-refractory; GVAX; Chemotherapy; Taxotere; Docetaxel; Prednisone; Vaccine; Allogeneic cells; Advanced Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Immunotherapy; Drug Therapy; Docetaxel; Prednisone

ARMS (2):
- 2 (Other): Standard of care - chemotherapy
  Interventions: Drug: Chemotherapy (Taxotere and prednisone)
- 1 (Experimental): Immunotherapy
  Interventions: Biological: Immunotherapy with allogeneic prostate vaccine

INTERVENTIONS:
Biological: Immunotherapy with allogeneic prostate vaccine — Immunotherapy with allogeneic prostate vaccine
  Arms: 1
Drug: Chemotherapy (Taxotere and prednisone) — Chemotherapy (Taxotere and prednisone)
  Arms: 2

SUMMARY:
The purpose of this study is to compare the duration of survival between GVAX® immunotherapy for prostate cancer and chemotherapy treatment in patients with prostate cancer who no longer respond to hormone therapy, who have documented metastases, and who have not been treated with chemotherapy in the past.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of or clinical history consistent with adenocarcinoma of the prostate
* Metastatic prostate cancer deemed to be unresponsive or refractory to hormone therapy
* Detectable metastases
* Any Gleason score
* ECOG performance status 0-2

Exclusion Criteria:

* Prior treatment with chemotherapy
* Prior Immunotherapy
* Prior treatment with gene therapy
* Significant cancer related pain

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2004-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Survival | 0

SECONDARY OUTCOMES:
Bone pain and bone related events | 0

CONTACTS AND LOCATIONS:
Locations (125):
- United States (82):
  - Central Alabama Oncology, LLC, Alabaster, Alabama
  - Alaska Clinical Research Center, Anchorage, Alaska
  - Palo Verde Hematology/Oncology, Glendale, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - ACRC/Arizona Clinical Res. Ctr. Inc., Tuscon, Arizona
  - Arkansas Cancer Research Center, Little Rock, Arkansas
  - Compassionate Cancer Care Medical Group, Inc., Corona, California
  - Pacific Coast Hem Onc. Medical Group, Fountain Valley, California
  - California Cancer Care, Greenbrae, California
  - Center for Urological Research, La Mesa, California
  - Oncology Care Medical Associates, Montebello, California
  - UC Irvine Medical Center, Orange, California
  - San Bernardino Urological Associates, San Bernardino, California
  - Sharp Healthcare, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Cancer Research & Prevention Center, Soquel, California
  - San Diego Cancer Center, Vista, California
  - Univ. of Colorado Health Science Center, Aurora, Colorado
  - Cancer Center of Colorado Springs, Colorado Springs, Colorado
  - The Hope Clinic, Bristol, Connecticut
  - Urology Center of Grove Hill, New Britain, Connecticut
  - Carl & Dorothy Bennett Cancer Center, Stamford, Connecticut
  - Boca Raton Community Hospital, Inc., Boca Raton, Florida
  - Michael and Dianne Bienes Comprehensive Cancer Center, Holy Cross Hospital, Fort Lauderdale, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Oncology-Hematology Group of South Florida/Advanced Medical Specialists, Miami, Florida
  - Cancer Centers of Florida, Ocoee, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Urology Consultants, Safety Harbor, Florida
  - Atlanta VAMC, Atlanta, Georgia
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Peachtree Hematology Oncology Consultants, PC, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Central Georgia Cancer Care, P.C., Macon, Georgia
  - Straub Clinic & Hospital, Honolulu, Hawaii
  - University of Illinois at Chicago, Chicago, Illinois
  - Welborn Clinic Research Center, Evansville, Indiana
  - Fort Wayne Medical Oncology/Hematology Inc., Fort Wayne, Indiana
  - Louisiana Oncology Associates, Lafayette, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - West Michigan Regional Cancer and Blood Center, Free Soil, Michigan
  - William Beaumont Hospital, Cancer Clinical Trials Office, Royal Oak, Michigan
  - Newland Medical Associates, P.C., Southfield, Michigan
  - Hematology Oncology Consultants, Inc., St Louis, Missouri
  - Deaconess Billings Clinic, Billings, Montana
  - Hematology/Oncology Centers of the Northern Rockies, P.C., Billings, Montana
  - Omaha VA Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - The Center for Cancer & Hematologic Disease, Cherry Hill, New Jersey
  - Hematology-Oncology Associates of Northern New Jersey, Morristown, New Jersey
  - Summit Medical Group/Overlook Oncology Center, Summit, New Jersey
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Jacobi Medical Center, The Bronx, New York
  - Presbyterian Hospital/ Center for Cancer Research, Charlotte, North Carolina
  - Northwestern Carolina Hematology Oncology, PA, Hickory, North Carolina
  - Medcenter One Cancer Care / Odyssey Research, Bismarck, North Dakota
  - Dakota Cancer Institute, Fargo, North Dakota
  - Gabrail Cancer Center, Canton, Ohio
  - Cleveland Clinic Foundation, Taussig Cancer Center, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Urologic Surgery PC, Bala-Cynwyd, Pennsylvania
  - Medical Oncology Associates, Kingston, Pennsylvania
  - Lancaster Cancer Center, Ltd, Lancaster, Pennsylvania
  - Urological Associates of Lancaster, Lancaster, Pennsylvania
  - University of Pittsburgh Cancer Center, Pittsburgh, Pennsylvania
  - Charleston Hematology Oncology, Charleston, South Carolina
  - Memorial Health Care System, Chattanooga, Tennessee
  - The West Clinic, Memphis, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Center for Oncology Research and Treatment PA, Dallas, Texas
  - Urology Specialists and Associates, P.A., Dallas, Texas
  - Mobley Research Center, Houston, Texas
  - Urology San Antonio, San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Southwestern Oncology Research Department, Bennington, Vermont
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Mason Medical Center Urology, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
- Belgium (9):
  - ZNA Middelheim, Antwerp
  - Imelda Ziekenhuis, Bonheiden
  - University Hospital Antwerp (UZA), Edegem
  - UZ Gent, Ghent
  - Unversity Hospial Gent, Ghent
  - Virga Jesse Ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk
  - Heilig Hartziekenhuis Roeselare Men, Roeselare
  - Regionaal Ziekenhuis Sint Trudo, Sint-Truiden
- Canada (5):
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUM Notre-Dam, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Ultra Med Inc., Pointe-Claire, Quebec
  - Centre Hopitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- France (8):
  - Centre Paul Papin, Angers
  - Centre Francois Baclesse, Caen
  - Centre Georges Francois Leclerc, Dijon
  - Centre Leon Berard Service de Cancerologie Medicale, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Centre Rene Gauducheau, Nantes-Saint Herblain
  - Institut Jean Godinot, Reims
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
- Germany (4):
  - Universitatsklinikum Aachen Urologie, Aachen
  - der Technischen Universitat Dresden, Dresden
  - Universitatsklinik um Essen, Essen
  - Universitatsklinik um des Saarlande, Homburg/Saar
- Netherlands (2):
  - VU Medisch Centrum, Amsterdam
  - University Medical Centre Groningen, Groningen
- Sweden (3):
  - University Hospital, Linkoping, Linköping
  - University Hospital Lund, Lund
  - Akademiska University Hospital, Uppsala
- United Kingdom (12):
  - Addenbrooke's Hospital, Cambridge
  - Beatson Oncology Centre, Glasgow
  - St. James's University Hospital, Leeds
  - Hammersmith Hospital, London
  - Mount Vernon Hospital, Middlesex
  - Newcastle General Hospital, Newcastle upon Tyne
  - Northampton General Hosptial, Northampton
  - Nottingham City Hospital, Nottingham
  - Oxford Cancer Centre, Churchill Hospital, Oxford
  - Scunthorpe General Hospital, Scunthorpe
  - Royal Hallamshire Hospital, Sheffield
  - Glan Clwyd Hospital, Wales

REFERENCES:
- [Derived] Vuky J, Corman JM, Porter C, Olgac S, Auerbach E, Dahl K. Phase II trial of neoadjuvant docetaxel and CG1940/CG8711 followed by radical prostatectomy in patients with high-risk clinically localized prostate cancer. Oncologist. 2013 Jun;18(6):687-8. doi: 10.1634/theoncologist.2011-0234. Epub 2013 Jun 5. PMID 23740935